CLINICAL TRIAL: NCT07335913
Title: A PHASE 1, TWO-PART, DOUBLE-BLIND, RANDOMIZED, PLACEBO CONTROLLED STUDY EVALUATING THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF SINGLE AND MULTIPLE ASCENDING DOSES OF ORALLY ADMINISTERED SBS-147 IN HEALTHY ADULTS
Brief Title: Phase 1 Study of SBS-147 in Healthy Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sparian Biosciences, Inc (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); Altasciences Company Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBS147-AP-107
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Pain Acute; Pain
Keywords: Arylepoxamide; AEAr Agonist; 6TM; Tolerability; Safety; SBS-147; SBS147
MeSH Terms: conditions — Acute Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (Experimental): Single dose of SBS-147 or a placebo given during trial
  Interventions: Drug: SBS-147; Drug: Placebo
- Multiple Ascending Dose (Experimental): SBS-147 or placebo given repeatedly over several days during the trial
  Interventions: Drug: SBS-147; Drug: Placebo

INTERVENTIONS:
Drug: SBS-147 — Experimental therapeutic
Drug: Placebo — Placebo comparator

SUMMARY:
This study is part of the HEAL Initiative supported by the NIH.

The purpose of this study is to learn how safe the study drug, SBS-147, is and how people's bodies respond to and process it. Researchers will also look for any side effects that may occur when taking SBS-147.

Some participants will receive SBS-147, and others will receive a placebo, which looks the same but does not contain any medicine. This helps researchers fairly compare results.

The study includes two parts:

Single-Dose Group, where Participants receive SBS-147 or placebo one time.

Multiple-Dose Group, where Participants receive SBS-147 or placebo once or twice daily for 7 days.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn about the safety of SBS-147. The main questions it aims to answer are:

What medical problems do participants have when taking SBS-147? Researchers will compare SBS-147 to a placebo (a look-alike substance that contains no drug) to see if SBS-147 works to treat acute pain.

Participants in the single ascending dose portion will:

Take SBS-147 or a placebo one time during the study Stay confined to the clinic for a period of 5 days and undergo tests, blood draws, and questionnaires.

Complete an end of study visit on Day 8

Participants in the multiple ascending dose portion will:

Take SBS-147 or a placebo one time per day or twice a day for 7 days Stay confined to the clinic for a period of 10 days and undergo tests, blood draws, and questionnaires.

Complete an end of study visit on Day 14

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF)
2. Healthy adult male or female, aged 18 to 55 years, inclusive, at Screening
3. Body mass index (BMI) within 18.0 kg/m2 to 32.0 kg/m2 inclusively
4. Minimum body weight of at least 50.0 kg at Screening
5. Stated willingness to comply with all study procedures and availability for the duration of the study
6. Females of childbearing potential
7. Healthy, as determined by protocol requirements
8. Non- or ex-smoker for at least 90 days prior to Screening
9. Participant is able and willing to comply with all study protocol procedures and requirements

Exclusion Criteria:

1. Female who is lactating at Screening
2. Female who is pregnant
3. History of significant hypersensitivity reactions (like angioedema) to any drugs
4. Presence or history of significant surgery that may affect drug bioavailability
5. History of significant CV, pulmonary, hematologic, neurologic, psychiatric, endocrine, infectious, or immunologic disease
6. Meet Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5) criteria for lifetime or current substance use disorder for any psychoactive substances other than nicotine or caffeine
7. Showing suicidal tendency as per the C-SSRS administered at screening and clinic admission
8. Any clinically significant illness in the 28 days prior to the first study drug administration
9. Use of any prescription drugs in the 28 days or 5 half-lives, whichever is longer, prior to Screening and until the end of the study, that in the opinion of an Investigator would put into question the status of the participant as healthy
10. Use of opioids, hypnotics, and/or sedatives in the last 30 days prior to screening
11. Routine or chronic use of acetaminophen or nonsteroidal anti-inflammatory drugs for more than 7 of the 20 days during the screening period.
12. Use of St. John's Wort in the 28 days prior to Screening
13. Use of any herbal supplements (including Kratom) the 14 days prior to Screening
14. Intake of an Investigational Product (IP) in the 30 days prior to Screening
15. Positive test result for alcohol and/or drugs of abuse at Screening or prior to the first drug administration
16. Positive screening results to HIV Ag/Ab combo, hepatitis B surface antigen or hepatitis C virus Ab tests
17. Any other clinically significant abnormalities in laboratory test results at screening that would, in the opinion of an Investigator and based on clinical judgment, increase the participant's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data
18. Donation of plasma in the 7 days prior to Screening
19. Donation of 1 unit of blood to American Red Cross or equivalent organization or donation of over 500 mL of blood in the 56 days prior to Screening
20. Inclusion in a previous cohort for this clinical study
21. Supine pulse rate less than 45 beats per minute (bpm) or more than 100 bpm at the screening visit
22. Supine systolic blood pressure < 90 or > 140 mmHg or diastolic blood pressure < 40 or > 90 mmHg at the Screening visit
23. Oxygen saturation (SpO2) below 95% at the Screening visit
24. Presence of out-of-range cardiac interval on the ECG at screening or other clinically significant ECG abnormalities, unless deemed non-significant by an Investigator
25. History of risk factors for Torsades de Pointes, including unexplained syncope, known long QT syndrome, heart failure, myocardial infarction, angina, or clinically significant abnormal laboratory assessments including hypokalaemia, hypercalcaemia, or hypomagnesaemia
26. Family history of long QT syndrome or Brugada syndrome
27. History of fainting
28. Family history of sudden cardiac death or significant heart disease
29. Known presence or history of gastroesophageal reflux or hiatal hernia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 8 days
  To assess the number of treatment emergent adverse events experienced in participants after a single dose of SBS-147
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 at ascending doses | 14 days
  Assess the number of treatment emergent adverse events experienced by participants of SBS-147 after multiple dose oral administration in healthy adults.

SECONDARY OUTCOMES:
Relative plasma exposure of SBS-1000 compared with SBS-147 (SAD) | 0-12 hours, 0-24 hours, and extrapolated to infinity after dosing
  Geometric mean ratios (SBS-1000 / SBS-147) for Cmax and AUC
Plasma pharmacokinetics of SBS-1000 and SBS-147 following multiple ascending doses | Day 1 (single-dose PK) and Day 7 at steady state over the dosing interval (τ)
  Plasma concentrations of SBS-1000 and SBS-147 will be analyzed using noncompartmental methods to characterize single-dose and steady-state pharmacokinetics.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Reich, MD, Study Director — Sparian Biosciences
Locations (1):
- AltaSciences, Inc, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No